CLINICAL TRIAL: NCT05343897
Title: Training Effects on Ping-Shuai-Gong and Arm-Swing-Exercise
Brief Title: Effects of Ping-Shuai-Gong and Arm-Swing-Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Fong Chin Su, Emeritus Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 109-490
Record Dates: First submitted 2021-10-25; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Effects of; Movement; Inactivity, Physical; Degeneration
Keywords: Ping Shuai Gong; Arm Swing Exercise; low intensity exercise; cardiovascular system; cerebrovascular system; microcirculatory blood flow; balance
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2-month Ping-Shuai Gong (PSG) training (Experimental): Ping-Shuai Gong (PSG) is pioneered by Qi Gong master, Li Feng-shan. It is featured in synchronous and rhythmic arm-swinging movement, with arms straightly forward flexing to shoulder level and backward extending repeatedly, and combined with lightly squat twice while arms swing to the fifth time and continue this cycle.
  They were asked to conduct and record 30 minutes of PSG in one day lasting for 2-month, and at least 3 days a week.
  Interventions: Behavioral: Low intensity exercise - Ping-Shuai Gong (PSG)
- 2-month Arm-Swing-Exercise (ASE) training (Active Comparator): Participents in Arm-Swing-Exercise (ASE) group were instructed to keep whole upper limbs pronated, and maintain their trunk straight while movement. The movement is to swing bilateral arms forward to around 30 degree and backward to around 60 degree continuously. The participants need to stabilize their trunk, pelvic, and legs while bilateral arms swinging passing through the side of the trunk. The most significant difference from PSG group is the way they pull the arm, not just swing backward and downward.
  They were asked to conduct and record 30 minutes of ASE in one day lasting for 2-month, and at least 3 days a week.
  Interventions: Behavioral: Low intensity exercise - Arm-Swing Exercise (ASE)

INTERVENTIONS:
Behavioral: Low intensity exercise - Ping-Shuai Gong (PSG) — Participants were asked to conduct and record 30 minutes of PSG in one day lasting for 2-month, and at least 3 days a week. A record sheet were sent to the participants in the first time, and the contact information of examiner were given as well. The examiner will check the completion of exercise execution via phone every two to three days and visit participants to confirm the correctness of movement at least one time during the 2-month intervention period.
  Arms: 2-month Ping-Shuai Gong (PSG) training
Behavioral: Low intensity exercise - Arm-Swing Exercise (ASE) — Participants were asked to conduct and record 30 minutes of ASE in one day lasting for 2-month, and at least 3 days a week. A record sheet were sent to the participants in the first time, and the contact information of examiner were given as well. The examiner will check the completion of exercise execution via phone every two to three days and visit participants to confirm the correctness of movement at least one time during the 2-month intervention period.
  Arms: 2-month Arm-Swing-Exercise (ASE) training

SUMMARY:
Ping Shuai Gong (PSG) and Arm Swing Exercise (ASE) are two similar exercise with different arm-swinging strategies. This study is plan to explore the relationship between characteristics of arm-swinging movement and skin blood flow during exercise.

DETAILED DESCRIPTION:
With the development of an aging society, the health and social systems of the elderly population have become issues that cannot be ignored. Due to the features of low difficulty and small space requirements, Ping Shuai Gong (PSG) and Arm Swing Exercise (ASE) become very popular within the older population. These physical activities have been proved to show advancement in cardiovascular and physical functions. Hence, this study is design to explores the health effects of two different arm-swinging strategies, and to explore the relationship between characteristics of arm-swinging movement and skin blood flow during exercise.

40 elderly people over 60 years old who have no regular exercise habits were divided into PSG group and ASE group, and each group was given two months of exercise training (at least 24 times of exercise, 30 minutes totally within one day). PSG group was asked to perform PSG exercises (actions were synchronized with the hands raised to shoulder height and then swinging down and back, with two squatting movements at the fifth time). ASE group was asked to perform ASE exercises (actions were to raise both hands synchronously to a 30-degree bend and then 60-degree shoulder extension, and to control the stability of the upper body when swinging arms).

Evaluation procedures of the pretraining evaluation and post-training evaluation are exactly the same.

ELIGIBILITY:
Inclusion Criteria:

age over 60 able to stand unassisted for at least 30 minutes able to understand and follow the instructions no good exercise habits (frequency > 3 times / wk.), intensity (rated perceived exertion > 12/20), time > 30 min.) for at least 3 months able to attend the experiment for 2 months

Exclusion Criteria:

uncontrolled cardiovascular disease severe arrhythmia peripheral artery disease respiratory system diseasehemodialysis patients unresolved upper or lower extremity injury

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-07-03 (Actual); Study Completion 2021-07-03 (Actual)

PRIMARY OUTCOMES:
cardiovascular system | 2 months
  Heart rate (HR), heart rate variability (HRV) to assess cardiac autonomic regulation.
cardiovascular system | 2 months
  blood pressue
cardiovascular system | 2 months
  Static photoplethysmography (PPG) signals were applied to measure low frequency oscillations of microvascular system, calculated as coefficient of variation (CV) of specific pulsation oscillation frequency, to assess vessel conditions for dynamic adaption in hemodynamics and biological signals. In each frequency interval, cardiac activity intensity is represented in 0.6 to 2 Hz oscillation and respiratory activity is from 0.145 to 0.6 Hz, myogenic activity is from 0.052 to 0.145 Hz, neurogenic activity is from 0.021 to 0.052 Hz, and NO-dependent endothelial activity is microvessel oscillation from 0.0095 to 0.021 Hz.

SECONDARY OUTCOMES:
cerebrovascular system | 2 months
  Changes in oxygenated (HbO) and deoxygenated (Hb) hemoglobin concentrations measured from NIRs to assess brain activation in motor-related cortex.
balance ability | 2 months
  Ground reaction force, rate of force development (RFD)/body weight , and total time in five-time sit to stand test (5XSST) measured from forceplates to assess strength.
balance ability | 2 months
  Center of pressure of five-time sit to stand test (5XSST) measured from forceplates to assess dynamic stability.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ping Shuai Gong video — https://www.youtube.com/watch?v=4nOIvWi4K_8&t=1s